CLINICAL TRIAL: NCT02754804
Title: Claudication et Fatigue Musculaire de l'artériopathe
Brief Title: Claudication, Systematic Evaluation of Limp on Treadmill
Acronym: CLAUSEL
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-A000052-49
Record Dates: First submitted 2016-04-16; First posted 2016-04-28 (Estimated); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PAD patients: Patients with grade 1 claudication Measurement of biomechanic parameters while walking on treadmill
  Interventions: Device: Biomechanic parameters

INTERVENTIONS:
Device: Biomechanic parameters — recording of biomechanic parameters and surface electromyography at the thigh and calf level throughout the walking period, in PAD patients .

SUMMARY:
Vascular claudication is a common cause of functional limitation. This painful condition is a source overall muscle deconditioning in the peripheral arterial diseased (PAD) patient leading gradually to a state accented inactivity. The characterization of the claudication as it results from a proximal or distal ischemia has never carried out. Investigators will analyze dynamic pedometer parameter throughout walking tests in PAD patients with claudication

DETAILED DESCRIPTION:
Patients referred for exercise tests on treadmill for the quantification of walking ability will gave a recording of their walking parameters through an instrumented treadmill recording biomechanic parameters (surface electromyography, walking pace; force of the foot/treadmill interface, length of the step.. etc.) Analysis will be performed until walking is stopped due to usual claudication during a constant load 2 miles per hour 10% slope treadmill procedure.

ELIGIBILITY:
Inclusion Criteria:

* Referred for treadmill testing
* Age > 18
* Claudication
* Covered by the French Healthcare system
* Consent to participate

Exclusion Criteria:

* Unstable angina
* History of lower limb osteo articular rheumatologic disease
* Lower limb amputation
* Cardiac or respiratory failure
* Neurologic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients complaining claudication and referred for a treadmill test
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2020-03-12 (Actual)

PRIMARY OUTCOMES:
Root mean square (RMS) of the electromyogram signal | Evaluation is complete immediately at the end of each walking test. (The end of the walking period is the end of participation of each patient, no follow up of patients)
  Calculation for the difference (change) in RMS value at the end vs.beginning of the walking test (RMS is calculated over 15 sec at rest and 15 sec just before the end of the walking period)

CONTACTS AND LOCATIONS:
Overall Officials: pierre Abraham, MD PhD, Principal Investigator — University Hospital, Angers
Locations (1):
- Centre hospitalier universitaire, Angers, France

IPD SHARING:
Plan to Share IPD: No